CLINICAL TRIAL: NCT02753595
Title: A Randomized, Open-label, Multicenter, Phase 1b/2 Study of Eribulin Mesylate in Combination With PEGylated Recombinant Human Hyaluronidase (PEGPH20) Versus Eribulin Mesylate Alone in Subjects With Human Epidermal Growth Factor Receptor 2 (HER2)-Negative, High-Hyaluronan (HA) Metastatic Breast Cancer (MBC)
Brief Title: Study of Eribulin Mesylate in Combination With PEGylated Recombinant Human Hyaluronidase (PEGPH20) Versus Eribulin Mesylate Alone in Subjects With Human Epidermal Growth Factor Receptor 2 (HER2)-Negative, High-Hyaluronan (HA) Metastatic Breast Cancer (MBC)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: evolving standard of care and difficulties of enrolling participants
Sponsor: Eisai Inc. (Industry)
Collaborators: Halozyme Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E7389-M000-219; 2015-004740-19 (EudraCT Number)
Record Dates: First submitted 2016-04-26; First posted 2016-04-28 (Estimated); Results first posted 2020-07-13 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-06

CONDITIONS: Metastatic Breast Cancer
Keywords: PEGylated Recombinant Human Hyaluronidase; Eribulin Mesylate; E7389; PEGPH20; Human Epidermal Growth Factor Receptor 2-Negative; High-Hyaluronan
MeSH Terms: conditions — Breast Neoplasms | interventions — eribulin; PEGPH20

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Eribulin mesylate plus PEGPH20 (Phase 1b) (Experimental): Recommended Phase 2 dose (RP2D) will be determined from the below dose levels:
  * Dose level 1: PEGPH20 (3.0 microgram per kilogram (mcg/kg)) followed by eribulin mesylate (1.4 milligrams per square meter (mg/m^2)) or
  * Dose level 0: PEGPH20 (1.6 mcg/kg) followed by eribulin mesylate (1.4 mg/m^2) or
  * Dose level -1: PEGPH20 (1.6 mcg/kg) followed by eribulin mesylate (1.1 mg/m^2)
  Dose level 1 can be selected as the RP2D if no more than 1 out of 6 participants has a DLT; DLT was only observed from the first treatment cycle; otherwise, Dose level 0 will be assessed in a second cohort of 6 subjects and will be selected as the RP2D if no more than 1 subject has a DLT. Otherwise, Dose level - 1 will be assessed in a third cohort of 6 subjects. Upon determination of the RP2D, study Phase 1b Expansion Part will proceed to confirm the RP2D, and thereafter Phase 2 part will proceed.
  Interventions: Drug: Eribulin mesylate; Other: Biologic: PEGylated recombinant human hyaluronidase (PEGPH20)
- Eribulin mesylate plus PEGPH20 (Phase 2) (Experimental): Participants will receive eribulin mesylate and PEGPH20 at the established RP2D level achieved in the Phase 1b.
  Interventions: Drug: Eribulin mesylate; Other: Biologic: PEGylated recombinant human hyaluronidase
- Eribulin mesylate (Phase 2) (Experimental): Participants will receive eribulin mesylate at 1.4 mg/m^2.
  Interventions: Drug: Eribulin mesylate

INTERVENTIONS:
Drug: Eribulin mesylate — Eribulin mesylate will be administered at 1.4 mg/m^2 or 1.1 mg/m^2 as intravenous (IV) infusion on Day 1 and 8 of 21-day cycle
  Other Names: E7389
  Arms: Eribulin mesylate plus PEGPH20 (Phase 1b)
Drug: Eribulin mesylate — Eribulin mesylate will be administered at 1.4 mg/m^2 or 1.1 mg/m^2, depending on RP2D, as IV infusion on Day 1 and 8 of each 21-day cycle
  Other Names: E7389
  Arms: Eribulin mesylate plus PEGPH20 (Phase 2)
Drug: Eribulin mesylate — Eribulin mesylate will be administered at 1.4 mg/m^2 as IV infusion on Day 1 and 8 of 21-day cycle
  Other Names: E7389
  Arms: Eribulin mesylate (Phase 2)
Other: Biologic: PEGylated recombinant human hyaluronidase (PEGPH20) — PEGPH20 will be administered at 3.0 mcg/kg or 1.6 mcg/kg as IV infusion on Day -1 and 7 of 21-day cycle
  Arms: Eribulin mesylate plus PEGPH20 (Phase 1b)
Other: Biologic: PEGylated recombinant human hyaluronidase — PEGPH20 will be administered at 3.0 mcg/kg or 1.6 mcg/kg, depending on RP2D, as IV infusion on Day -1 and 7 of each 21-day cycle
  Arms: Eribulin mesylate plus PEGPH20 (Phase 2)

SUMMARY:
The primary objective for the study is as follows:

For the Phase 1b - to determine safety tolerability and recommended Phase 2 dose (RP2D) of eribulin mesylate in combination with PEGylated recombinant human hyaluronidase (PEGPH20) in participants with Human Epidermal Growth Factor Receptor (HER2)-negative metastatic breast cancer (MBC) previously treated with up to two lines of systemic anticancer therapy in the metastatic setting.

For the Phase 2 - to evaluate objective response rate (ORR) of eribulin mesylate in combination with PEGPH20 in participants with HER2-negative, High-Hyaluronan (HA)-high, MBC previously treated with up to 2 lines of systemic anticancer therapy in the metastatic setting.

DETAILED DESCRIPTION:
Phase 1b will occur in two parts:

Part 1: Run-in safety cohort(s) (dose levels 1, 0, and -1, as necessary) of 6 participants each will be conducted until the RP2D is determined. The purpose of the run-in safety cohort(s) is to study the safety of the 2-drug combination and determine a RP2D. Dose limiting toxicity (DLT) will be assessed in the first cycle to determine the RP2D of eribulin mesylate in combination with PEGPH20.

Part 2 (Phase 1b "Expansion Part"): A total of 12 additional participants will be enrolled at the RP2D determined in Part 1 (using Phase 1b criteria, i.e., participants previously treated with up to 2 lines of systemic anticancer therapy) in order to assess the safety profile of the combination and identify any potential safety signals and the incidence of thromboembolic events in this population (RP2D determined dosing).

In Phase 2, participants will be stratified by triple negative breast cancer (TNBC) status and randomized 1:1 to receive eribulin mesylate and PEGPH20 at the established RP2D level or eribulin mesylate alone at 1.4 milligrams per square meters (mg/m^2).

ELIGIBILITY:
Inclusion Criteria

1. Metastatic Her-2- breast cancer
2. Up to 2 prior lines of cytotoxic or targeted anti-cancer therapy for metastatic disease
3. Measurable disease per Response Evaluation Criteria In Solid Tumors (RECIST) v1.1
4. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1

Exclusion Criteria

1. Less than 6 months since prior neoadjuvant/adjuvant chemotherapy
2. Known central nervous system (CNS) disease, except for those participants with treated brain metastasis who are stable for at least 1 month, having no evidence of progression or hemorrhage after treatment and no ongoing requirement for corticosteroids, as ascertained by clinical examination and brain imaging (MRI or CT) during the screening period
3. Previous history or current evidence of deep vein thrombosis (DVT), hereditary thrombophilic syndromes, pulmonary embolism (PE), cerebral vascular accident (CVA), transient ischemic attack (TIA), atrial fibrillation (AF), or active carotid artery disease requiring treatment
4. Treatment with chemotherapy, hormonal, or biological therapy within the previous 3 weeks, radiation or small molecule targeted therapy within the previous 2 weeks preceding informed consent
5. Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-07-13 (Actual); Primary Completion 2019-08-16 (Actual); Study Completion 2019-08-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Whittier, California
  - Atlanta, Georgia
  - Newnan, Georgia
  - Anderson, Indiana
  - Bethesda, Maryland
  - Stony Brook, New York
  - Kennewick, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 4 investigative sites in the United States from 13 Jul 2016 to 16 Aug 2019. A total of 25 participants were screened and enrolled (signed informed consent form), of which 11 were screen failures, and 14 were treated.
Pre-assignment Details: Study terminated early during Phase 1b Expansion Part and before initiating Phase 2 due to poor accrual. Data reported is based on initial dosing levels given to participants during Phase 1b. Combined data for participants who received Dose level 0 during determination of RP2D and confirmation of RP2D (Expansion Part) are reported as planned.
Groups:
- Phase 1b: Dose Level 1: Participants received PEGylated recombinant human hyaluronidase (PEGPH20) 3.0 microgram per kilogram (mcg/kg), infusion, intravenously on Days -1 and 7 followed by eribulin mesylate 1.4 milligram per square meter (mg/m^2), infusion, intravenously, on Days 1 and 8 of each 21-day treatment cycle up to Cycle 28 (Dose level 1).
- Phase 1b: Dose Level 0 and Expansion Part: Participants received PEGPH20 1.6 mcg/kg, infusion, intravenously on Days -1 and 7 followed by eribulin mesylate 1.4 mg/m^2, infusion, intravenously, on Days 1 and 8 of each 21-day treatment cycle for up to Cycle 28 (Dose Level 0). After the determination of RP2D at this dosing level in Cycle 1 of Phase 1b, additional participants were enrolled in this dosing level for the confirmation of the RP2D in the Expansion Part for up to Cycle 28.
Period: Overall Study
Arm/Group | Phase 1b: Dose Level 1 | Phase 1b: Dose Level 0 and Expansion Part
Started | 5 | 9
Completed | 3 | 7
Not Completed | 2 | 2
Not completed — Sponsor termination | 2 | 2

BASELINE CHARACTERISTICS:
Population: The safety analysis set included participants who received at least 1 dose of the study drug in Phase 1b.
Groups:
- Phase 1b: Dose Level 1: Participants received PEGPH20 3.0 mcg/kg, infusion, intravenously on Days -1 and 7 followed by eribulin mesylate 1.4 mg/m^2, infusion, intravenously, on Days 1 and 8 of each 21-day treatment cycle up to Cycle 28 (Dose level 1).
- Total: Total of all reporting groups
Arm/Group | Phase 1b: Dose Level 1 | Phase 1b: Dose Level 0 and Expansion Part | Total
Number analyzed (Participants) | 5 | 9 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.2 (13.10) | 52.8 (11.86) | 53.6 (11.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 9 | 14
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3
  Not Hispanic or Latino | 5 | 6 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 2 | 4 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 4 | 4

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b: Recommended Phase 2 Dose (RP2D) of Eribulin Mesylate in Combination With PEGPH20
Description: The RP2D was the maximum tolerated dose (MTD) or less. The MTD was determined as the dose level (1, 0) at which less than or equal to (<=) 1 of 6 evaluable participants experienced dose limiting toxicity (DLT) within the first 21 days of treatment (end of Cycle 1). Upon determination of RP2D in Cycle 1 of Phase 1b, RP2D was to be confirmed in Phase 1b-expansion Part.
Time Frame: Up to Cycle 28 (Cycle Length= 21 days)
Population: The safety analysis set included participants who received at least 1 dose of the study drug in Phase 1b.
Measure: Number; unit: mg/m^2
Groups:
- Phase 1b, All Participants: Participants received PEGPH20 3.0 mcg/kg or 1.6 mcg/kg, infusion, intravenously on Days -1 and 7 followed by eribulin mesylate 1.4 mg/m^2, infusion, intravenously, on Days 1 and 8 of first 21-day treatment cycle. After the determination of RP2D in Cycle 1 of Phase 1b, additional participants were enrolled for the confirmation of the RP2D in the Expansion Part for up to Cycle 28.
Arm/Group | Phase 1b, All Participants
Number analyzed (Participants) | 14
mg/m^2 | NA — RP2D was not confirmed due to early termination of study because of poor accrual before completing Phase 1b-expansion Part (which was planned for confirming the RP2D)

2. Primary Outcome: Phase 1b: Recommended Phase 2 Dose (RP2D) of PEGPH20 in Combination With Eribulin Mesylate
Description: The RP2D was the MTD or less. The MTD was determined as the dose level (1, 0) at which <=1 of 6 evaluable participants experienced DLT within the first 21 days of treatment (end of Cycle 1). Upon determination of RP2D in Cycle 1 of Phase 1b, RP2D was to be confirmed in Phase 1b-expansion Part.
Time Frame: Up to Cycle 28 (Cycle Length= 21 days)
Population: The safety analysis set included participants who received at least 1 dose of the study drug in Phase 1b.
Measure: Number; unit: mcg/kg
Arm/Group | Phase 1b, All Participants
Number analyzed (Participants) | 14
mcg/kg | NA — RP2D was not confirmed due to early termination of study because of poor accrual before completing Phase 1b-expansion Part (which was planned for confirming the RP2D)

ADVERSE EVENTS:
Time Frame: From the first dose of study drug up to approximately 3 years 1 month
Description: Deaths that happened anytime during the study (including those during the treatment and after treatment discontinuation) are reported in this section.
Arm/Group | Phase 1b: Dose Level 1 | Phase 1b: Dose Level 0 and Expansion Part
All-Cause Mortality (participants affected / at risk) | 2/5 | 3/9
Serious Adverse Events (participants affected / at risk) | 1/5 | 3/9
Other Adverse Events (participants affected / at risk) | 5/5 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b: Dose Level 1 (N=5) | Phase 1b: Dose Level 0 and Expansion Part (N=9)
Non-cardiac chest pain (General disorders) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pericardial effusion malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b: Dose Level 1 (N=5) | Phase 1b: Dose Level 0 and Expansion Part (N=9)
Anaemia (Blood and lymphatic system disorders) | 1 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 5
Vision blurred (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 3
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Catheter site inflammation (General disorders) | 0 | 1
Fatigue (General disorders) | 3 | 2
Nodule (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 3 | 2
Pain (General disorders) | 0 | 2
Peripheral swelling (General disorders) | 2 | 1
Ear infection (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 1
Scar (Injury, poisoning and procedural complications) | 0 | 1
Blood lactic acid increased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 2 | 2
Weight decreased (Investigations) | 1 | 0
White blood cell count decreased (Investigations) | 1 | 2
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 6
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 2 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Neurotoxicity (Nervous system disorders) | 2 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 1
Nocturia (Renal and urinary disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 1
Polyuria (Renal and urinary disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1
Breast pain (Reproductive system and breast disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
Scar pain (Skin and subcutaneous tissue disorders) | 0 | 1
Hot flush (Vascular disorders) | 0 | 1
Taste disorder (Nervous system disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Eye contusion (Injury, poisoning and procedural complications) | 0 | 1
Malaise (General disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
The outcome measures assessing efficacy are not applicable for results disclosure due to immaturity of the data, as the study was terminated early in Phase 1b-Expansion part and prior to the initiation and enrollment of Phase 2.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-10-27): https://cdn.clinicaltrials.gov/large-docs/95/NCT02753595/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-07): https://cdn.clinicaltrials.gov/large-docs/95/NCT02753595/SAP_001.pdf